CLINICAL TRIAL: NCT02852850
Title: In Vivo Molecular Imaging With Infliximab Antibody With FITC Predicts Therapeutic Response in Ulcerative Colitis
Brief Title: In Vivo Molecular Imaging Predicts Therapeutic Response in Ulcerative Colitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2016SDU-QILU-12
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Molecular Imaging With IFX-FITC: Endoscopic examination with the fluorescent antibody (IFX-FITC) was performed in patients with active ulcerative colitis before infliximab therapy was initiated. Labeled infliximab was applied topically via a standard spray catheter onto the most inflamed region of the bowel during colonoscopy, followed by CLE. In vivo imaging of inflamed areas of the intestinal mucosa showed a specific fluorescence signal of mTNF+ cells after topical application of labeled adalimumab. These specific fluorescence signals were recorded.

SUMMARY:
Molecular imaging with infliximab antibody with FITC has the potential to predict therapeutic responses to infliximab antibody and can be used for personalized medicine in ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active ulcerative colitis will receive infliximab antibody therapy.

Exclusion Criteria:

* Patients with impaired blood clotting.
* Patients with short bowel syndrome.
* Patients during the pregnancy and lactation period.
* Patients received enema therapy within 1 month before inclusion in the study, or had anti-TNF therapy within the last 12 months.
* Patients participated in another clinical trial or administrated other investigational drugs within 4 months prior to the screening visit.
* Patients with moderate to severe heart failure, active tuberculosis or acute infections.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active ulcerative colitis will receive infliximab antibody therapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The number of specific fluorescence signal of mTNF+ cells in patients with UC | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD,PHD, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China